CLINICAL TRIAL: NCT01509183
Title: Effectiveness of the Propeller Health (Formerly Asthmapolis) Monitoring System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reciprocal Labs (Industry)
Collaborators: California HealthCare Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-10
Record Dates: First submitted 2012-01-09; First posted 2012-01-12 (Estimated); Results first posted 2018-02-13 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Asthma
Keywords: asthma; healthcare utilization costs
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Active Comparator): Intervention group (IG) participants received access to and feedback from the Propeller Health System (formerly Asthmapolis System).
  Interventions: Device: Propeller Health System (formerly Asthmapolis System)
- Control Group (No Intervention): Control group (CG) participants were outfitted with sensors from the Propeller Health System, but did not receive feedback.

INTERVENTIONS:
Device: Propeller Health System (formerly Asthmapolis System) — The Propeller (formerly Asthmapolis) system works through the provision of information to patients and their providers. With the Propeller (formerly Asthmapolis) device in place, each actuation of a patient's rescue inhaler is recorded with an automatic time stamp; in many circumstances, the location at which the device is actuated is also captured and recorded. Actuation data are then securely transmitted to Propeller (formerly Asthmapolis) where events and an assessment of asthma control can be viewed in secure online interfaces. The information is also compiled into individual reports that are returned to the patient and his or her provider. Patients also receive customized suggestions for asthma management based on their actuation history.
  Arms: Intervention Group

SUMMARY:
Propeller Health is collaborating with Dignity Health (formerly Catholic Healthcare West (CHW)) to carry out a focused demonstration project to evaluate the effectiveness and potential cost savings of a deployment of the Propeller Health approach to asthma management. The Propeller Health goal is to bring together the best technology and asthma insight in order to provide Dignity Health with an engaging, data-driven chronic care program to improve asthma management and lower healthcare utilization costs, and to respond to prevention-focused reforms to health insurance laws.

This project has been designed to implement and evaluate a data-driven program to improve asthma management and control and lower direct costs through reductions in healthcare utilization. This program has been developed by Propeller Health and has gone through preliminary testing. Each subject participating in the study will receive an Propeller Health device, which captures the time and location of use of inhaled short-acting bronchodilators over a twelve-month period. This information is processed and delivered at regular intervals to the patient and his or her provider to support improved asthma management.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the impact of the adoption of the Propeller Health system into a healthcare organization, and to provide sufficient information to inform decision making for potential future adopters. The researchers believe that the Propeller Health system has the potential to improve asthma control by providing rescue inhaler actuation data and tailored asthma management tips to patients with uncontrolled asthma, and rescue inhaler actuation data to their providers. Improvements in asthma control should be reflected in reductions in healthcare utilization for asthma, and potentially for general healthcare utilization. Reductions in utilization would result in lower healthcare costs. The study has been designed to capture data on individual subject asthma control, and changes in utilization and costs over a one-year introduction period.

ELIGIBILITY:
Inclusion Criteria:

* Provider diagnosis of asthma (ICD9 493.xx);
* At least one healthcare utilization event in CHW within last 12 months; and
* Prescription for Short Acting Beta Agonist (SABA) at study intake.

Exclusion Criteria:

* Subject is under the age of 5 at the beginning of the study;
* Subject does not speak either English or Spanish;
* Subject does not have access to the Internet or email to receive reports; and
* Subject has substantial co-morbidity (provider diagnosis of COPD

Ages: 5 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2012-04; Primary Completion 2014-10 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajan K Merchant, MD, Principal Investigator — Catholic Healthcare West Medical Foundation
Locations (1):
- Woodland Medical Center, Woodland, California, United States

REFERENCES:
- [Result] Merchant RK, Inamdar R, Quade RC. Effectiveness of Population Health Management Using the Propeller Health Asthma Platform: A Randomized Clinical Trial. J Allergy Clin Immunol Pract. 2016 May-Jun;4(3):455-63. doi: 10.1016/j.jaip.2015.11.022. Epub 2016 Jan 8. PMID 26778246
- See also: Publication — https://pubmed.ncbi.nlm.nih.gov/26778246/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between April 2012 & June 2013 via an asthma registry, community outreach efforts, and provider referrals.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 250 | 245
Completed | 141 | 134
Not Completed | 109 | 111

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 250 | 245 | 495
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 74 | 75 | 149
  Between 18 and 65 years | 163 | 158 | 321
  >=65 years | 13 | 12 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 140 | 285
  Male | 105 | 105 | 210

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean SABA Use
Description: Mean SABA use as measured by the Propeller Health sensor during the period of intervention (12 months).
Time Frame: Change in mean SABA use over the course of 12 months
Measure: Mean (Standard Deviation); unit: mean puffs per day
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 250 | 245
mean puffs per day | -0.41 (0.69) | -0.31 (0.75)

2. Secondary Outcome: Change in the Proportion of SABA-free Days From Baseline to 12 Months
Description: Evaluate the change in the proportion of SABA-free days from baseline to 12 months
Time Frame: Baseline to 12 months
Measure: Number; unit: % Change in proportion of SABA-free days
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 250 | 245
% Change in proportion of SABA-free days | 21 | 17

ADVERSE EVENTS:
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/250 | 0/245
Serious Adverse Events (participants affected / at risk) | 0/250 | 0/245
Other Adverse Events (participants affected / at risk) | 0/250 | 0/245

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No